CLINICAL TRIAL: NCT04405505
Title: A Randomized, Positive Parallel Controlled, Multicenter Phase III Study of TQB2450 Injection Combined With Anlotinib Hydrochloride Capsule Versus Paclitaxel for Injection (Albumin Bound) in Subjects With Triple Negative Breast Cancer (TNBC)
Brief Title: A Study of TQB2450 Injection Combined With Anlotinib Hydrochloride Capsule Versus Paclitaxel for Injection (Albumin Bound) in Subjects With Triple Negative Breast Cancer (TNBC)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TQB2450-III-06
Record Dates: First submitted 2020-05-24; First posted 2020-05-28 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — anlotinib; Paclitaxel; Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQB2450 + Anlotinib (Experimental): TQB2450 1200 mg administered intravenously (IV) on Day 1 of each 21-day cycle ,Anlotinib capsules 12 mg given orally, once daily in 21-day cycle (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21).
  Interventions: Drug: TQB2450; Drug: Anlotinib
- Paclitaxel for injection (albumin bound) (Active Comparator): Paclitaxel for Injection (albumin bound) 100mg / m2 administered intravenously (IV) on Day 1, 8, 15 in 28-day cycle.
  Interventions: Drug: Paclitaxel for Injection (albumin bound)

INTERVENTIONS:
Drug: TQB2450 — TQB2450 is a humanized monoclonal antibody targeting programmed death ligand-1 (PD-L1), which prevents PD-L1 from binding to PD-1 and B7.1 receptors on T cell surface, restores T cell activity, thus enhancing immune response and has potential to treat various types of tumors.
  Arms: TQB2450 + Anlotinib
Drug: Anlotinib — a multi-target receptor tyrosine kinase inhibitor.
  Arms: TQB2450 + Anlotinib
Drug: Paclitaxel for Injection (albumin bound) — a anti-microtubule drug.
  Arms: Paclitaxel for injection (albumin bound)

SUMMARY:
This study is a randomized, positive parallel controlled, multicentre phase III clinical trial to evaluate the efficacy and safety of TQB2450 combined with anlotinib versus paclitaxel for injection (albumin bound) in subjects with advanced triple negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1.Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1; Life expectancy ≥ 3 months.

  2.Histologically confirmed triple negative breast cancer. 3.Has at least one measurable lesion. 4.Newly diagnosed stage IV or recurrent/metastatic triple negative breast cancer who are not suitable for surgery.

  5.Prior local radiotherapy for metastatic sites is allowed. 6.Adequate laboratory indicators. 7.Understood and signed an informed consent form. 8.No pregnant or breastfeeding women, and a negative pregnancy test.

Exclusion Criteria:

* 1.Has received anti-angiogenic drugs or other PD-1 / PD-L1 / CTLA-4 antibody therapy or other immunotherapy against PD-1 / PD-L1 / CTLA-4.

  2. Severe hypersensitivity occurs after administration of other monoclonal antibodies.

  3. Has other malignancies (except cured skin basal cell carcinoma and cervical carcinoma in situ) within 3 years.

  4. Has any active autoimmune disease or history of autoimmune disease. 5. Has a clear clinical diagnosis of interstitial pneumonia, pulmonary fibrosis, drug-induced pneumonia, or active pneumonia.

  6. Peripheral neuropathy ≥ grade 2. 7. Immunosuppressant or systemic or absorbable local hormone therapy is required to achieve the aim of immunosuppression (dose > 10mg/ day prednisone or other therapeutic hormones) and is still used within 2 weeks after the first administration.

  8. Has multiple factors affecting oral medication. 9. Has uncontrolled and repeated drainage pleural effusion, pericardial effusion, and ascites.

  10. Has any signs of bleeding or history. 11. Has unrelieved spinal cord compression. 12. Has symptomatic central nervous system (CNS) disease and / or cancerous meningitis, pia mater disease.

  13. Has received other anti-tumor therapy within 4 weeks before the first administration.

  14. Has any serious and/or uncontrollable disease. 15. Has received vaccination or attenuated vaccine within 4 weeks before the first administration.

  16. According to the judgement of the investigators, there are other factors that may lead to the termination of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) evaluated by Independent Review Committee(IRC) | up to 96 weeks
  PFS defined as the time from randomization until the first documented progressive disease (PD) or death from any cause, based on IRC.

SECONDARY OUTCOMES:
Overall response rate (ORR) | up to 96 weeks
  Percentage of participants achieving complete response (CR) and partial response (PR).
Disease control rate（DCR） | up to 96 weeks
  Percentage of participants achieving complete response (CR) and partial response (PR) and stable disease (SD).
Duration of Response (DOR) | up to 96 weeks
  DOR defined as time from earliest date of disease response to earliest date of disease progression based on radiographic assessment.

CONTACTS AND LOCATIONS:
Locations (30):
- China (30):
  - The Fourth Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Chinese Academy of Medical Sciencesand Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Beijing Shijitan Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality
  - Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality
  - Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - The First Affilited Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Guangxi Medical University Affiliated Tumor Hospital, Nanning, Guangxi
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - The fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Affiliated Tumor Hospital of Harbin Medical University, Harbin, Heilongjiang
  - AnYang Tumor Hospital, Anyang, Henan
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Nantong Tumor Hospital, Nantong, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - Yanbian University Hospital, Yanji, Jilin
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - The Second Affiliated Hospital of PLA Airforce Military Medical University, Xi’an, Shanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Shanxi Provincial People's Hospital, Xi’an, Shanxi
  - The Second People's Hospital of Neijiang, Neijiang, Sichuan
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - Xinjiang Uiger Municipal People's Hospital, Ürümqi, Xinjiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang